CLINICAL TRIAL: NCT03563209
Title: Assesment of Post-stroke Elbow Flexor Spasticity in Response to Passive Stretch in Different Forearm Positions
Brief Title: Assesment of Post-stroke Elbow Flexor Spasticity in Different Forearm Positions
Status: Completed | Type: Observational
Sponsor: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, ilker şengül, Principal Investigator, Izmir Katip Celebi University
Other Study IDs: 21.02.2018-84
Record Dates: First submitted 2018-06-06; First posted 2018-06-20 (Actual); Results first posted 2019-05-10 (Actual); Last update posted 2019-05-22 (Actual); Status verified 2019-05

CONDITIONS: Post-stroke Elbow Spasticity
Keywords: Elbow spasticity; Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Determination of which muscle is more spastic before injection of the botulinum toxin, and the application of the targeted treatment to that muscle results in more improvement in spasticity. It is known that the muscles that flex elbow in healthy individuals change according to forearm position. While the biceps brachii flexes the forearm in supination, the brachioradialis flexes the forearm in the neutral position. The brachialis muscle acts as a primary flexor muscle when the forearm is in pronation.

In this study, hypothesis is that the severity of spasticity differs depending on the forearm position.

DETAILED DESCRIPTION:
There are three main muscles that contribute to elbow flexor spasticity; musculus biceps brachii, musculus brachialis and musculus brachioradialis. Muscle selection in elbow flexor spasticity for botulinum toxin application has impact on treatment outcome. The superficiality of the biceps brachii muscle makes it an easy target for botulinum toxin injection. In dynamic electromyography studies, it has been reported that brachioradialis muscle is the most common contributor one to elbow flexion spasticity, followed by biceps brachii muscle. In the diagnostic selective nerve blocks, the brachialis muscle has been reported to be foreground.

Determination of which muscle is more spastic before injection of the botulinum toxin, and the application of the targeted treatment to that muscle results in more improvement in spasticity. Can the target muscle selection clinically be performed instead of methods such as electromyography where equipment is required and the evaluation period is relatively long? Can semi-quantitative methods used to assess the severity of spasticity provide reliable information regarding the muscle or muscles that contribute to elbow flexor spasticity? It is known that the muscles that flex elbow in healthy individuals change according to forearm position. While the biceps brachii flexes the forearm in supination, the brachioradialis flexes the forearm in the neutral position. The brachialis muscle acts as a primary flexor muscle when the forearm is in pronation.

The aim of this study is to investigate whether the severity of spasticity differs depending on the forearm position.

ELIGIBILITY:
Inclusion Criteria:

* Elbow flexor spasticity
* Grade 1 to 3 spasticity measured with Modified Ashworth Scale
* To agree to participate in the study

Exclusion Criteria:

* <18 years old
* Pregnancy
* Botulinum toxin injection within the last three months
* Presence of elbow contracture
* History of operation to spastic upper extremity
* Spasticity due to other causes other than stroke
* Do not agree to participate in the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with post-stroke elbow flexor spasticity
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2018-03-15 (Actual); Primary Completion 2018-08-15 (Actual); Study Completion 2018-08-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ilker şengül, Principal Investigator — İzmir Katip Çelebi University
Locations (1):
- Ilker Şengül, Izmir, In the USA Or Canada, Please Select..., Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Keenan MA. Management of the spastic upper extremity in the neurologically impaired adult. Clin Orthop Relat Res. 1988 Aug;(233):116-25. PMID 3042230
- [Background] Genet F, Schnitzler A, Droz-Bartholet F, Salga M, Tatu L, Debaud C, Denormandie P, Parratte B. Successive motor nerve blocks to identify the muscles causing a spasticity pattern: example of the arm flexion pattern. J Anat. 2017 Jan;230(1):106-116. doi: 10.1111/joa.12538. Epub 2016 Sep 6. PMID 27595994
- [Background] Keenan MA, Haider TT, Stone LR. Dynamic electromyography to assess elbow spasticity. J Hand Surg Am. 1990 Jul;15(4):607-14. doi: 10.1016/s0363-5023(09)90023-5. PMID 2380525
- [Background] BASMAJIAN JV, LATIF A. Integrated actions and functions of the chief flexors of the elbow: a detailed electromyographic analysis. J Bone Joint Surg Am. 1957 Oct;39-A(5):1106-18. No abstract available. PMID 13475410
- [Background] Bohannon RW, Smith MB. Interrater reliability of a modified Ashworth scale of muscle spasticity. Phys Ther. 1987 Feb;67(2):206-7. doi: 10.1093/ptj/67.2.206. PMID 3809245
- [Background] Gracies JM, Bayle N, Vinti M, Alkandari S, Vu P, Loche CM, Colas C. Five-step clinical assessment in spastic paresis. Eur J Phys Rehabil Med. 2010 Sep;46(3):411-21. PMID 20927007

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study enrolled patients with post-stroke elbow flexor spasticity from a single medical center in Turkey. The last patients completed in July 2018
Groups:
- Post-stroke Elbow Flexor Spasticity: Participants with post-stroke elbow flexor spasticity
Period: Overall Study
Arm/Group | Post-stroke Elbow Flexor Spasticity
Started | 60
Completed | 60
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Post-stroke Elbow Flexor Spasticity
Number analyzed (Participants) | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 42
  >=65 years | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.82 (12.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 41
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 60
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Turkey | 60
Type of stroke [Count of Participants; unit: Participants]
  Ischemic | 45
  Hemoragic | 15
Side of plegia [Count of Participants; unit: Participants]
  Right | 26
  Left | 34
Disease duration [Median (Inter-Quartile Range); unit: months] | 38 [15.25 to 83.5]
Brunnstrom stage of motor recovery of upper extremity [Median (Inter-Quartile Range); unit: units on a scale] — The Brunnstrom recovery stages approach contains 3 subgroups (arm, hand and limb) which are scored separately on a 7-level likert scale (level I to VII).The stage I represents flaccid paralysis. Stage II marks the development of some synergy patterns. Spasticity reaches its peak in stage III. Spasticity begins to decrease in stage IV and patients have some normal movement patterns. In stage V, spasticity continues to decrease, and voluntary movements are more coordinated. In stage VI, motor control of the affected extremity is almost complete. Stage VII represents the return of full function.
  units on a scale | 3 [3 to 3]
Brunnstrom stage of motor recovery of hand [Mean (Inter-Quartile Range); unit: units on a scale] — The Brunnstrom recovery stages approach contains 3 subgroups (arm, hand and limb) which are scored separately on a 7-level likert scale (level I to VII).The stage I represents flaccid paralysis. Stage II marks the development of some synergy patterns. Spasticity reaches its peak in stage III. Spasticity begins to decrease in stage IV and patients have some normal movement patterns. In stage V, spasticity continues to decrease, and voluntary movements are more coordinated. In stage VI, motor control of the affected extremity is almost complete. Stage VII represents the return of full function.
  units on a scale | 3 [2 to 3]
Brunnstrom stage of motor recovery of lower extremity [Median (Inter-Quartile Range); unit: units on a scale] — The Brunnstrom recovery stages approach contains 3 subgroups (arm, hand and limb) which are scored separately on a 7-level likert scale (level I to VII).The stage I represents flaccid paralysis. Stage II marks the development of some synergy patterns. Spasticity reaches its peak in stage III. Spasticity begins to decrease in stage IV and patients have some normal movement patterns. In stage V, spasticity continues to decrease, and voluntary movements are more coordinated. In stage VI, motor control of the affected extremity is almost complete. Stage VII represents the return of full function.
  units on a scale | 3 [3 to 4]
Severity of spasticity according to the Modified Ashworth Scale in forearm pronation [Median (Inter-Quartile Range); unit: units on a scale] — The Modified Ashworth Scale indicates presence and severity of muscle spasticity. The Modified Ashworth Scale has 6 stages ranging between 0 to 4 (0, 1, 1+, 2, 3, 4). The severity of spasticity increases as the score increases. Score 0 represents no increase in tone, and in score 4, affected part is rigid. In statistical analysis, 6 stages ranging between 0 to 5 (0, 1, 2, 3, 4, 5) was used. Score of 1+ was treated as 2, 2 was treated as 3, 3 was treated as 4, and 4 was treated as 5.
  units on a scale | 3 [2 to 4]
Severity of spasticity according to the Modified Ashworth Scale in the neutral position of forearm [Median (Inter-Quartile Range); unit: units on a scale] — The Modified Ashworth Scale indicates presence and severity of muscle spasticity. The Modified Ashworth Scale has 6 stages ranging between 0 to 4 (0, 1, 1+, 2, 3, 4). The severity of spasticity increases as the score increases. Score 0 represents no increase in tone, and in score 4, affected part is rigid. In statistical analysis, 6 stages ranging between 0 to 5 (0, 1, 2, 3, 4, 5) was used. Score of 1+ was treated as 2, 2 was treated as 3, 3 was treated as 4, and 4 was treated as 5.
  units on a scale | 3 [2 to 4]
Severity of spasticity according to the Modified Ashworth Scale in forearm supination [Median (Inter-Quartile Range); unit: units on a scale] — The Modified Ashworth Scale indicates presence and severity of muscle spasticity. The Modified Ashworth Scale has 6 stages ranging between 0 to 4 (0, 1, 1+, 2, 3, 4). The severity of spasticity increases as the score increases. Score 0 represents no increase in tone, and in score 4, affected part is rigid. In statistical analysis, 6 stages ranging between 0 to 5 (0, 1, 2, 3, 4, 5) was used. Score of 1+ was treated as 2, 2 was treated as 3, 3 was treated as 4, and 4 was treated as 5.
  units on a scale | 3 [2 to 4]
Spontaneous elbow angle [Mean (Standard Deviation); unit: degree] | 118.17 (23.09)
Slow controlled motion (passive range of motion) of elbow joint in pronation [Median (Inter-Quartile Range); unit: degree] | 180 [180 to 180]
Slow controlled motion (passive range of motion) of elbow joint in the neutral position of forearm [Median (Inter-Quartile Range); unit: degree] | 180 [180 to 180]
Slow controlled motion (passive range of motion) of elbow joint in supination [Median (Inter-Quartile Range); unit: degree] | 180 [180 to 180]
Angle of muscle reaction in pronation [Median (Inter-Quartile Range); unit: degree] | 110 [100 to 123.75]
Angle of muscle reaction in the neutral position [Median (Inter-Quartile Range); unit: degree] | 115 [101.25 to 130]
Angle of muscle reaction in supination [Median (Inter-Quartile Range); unit: degree] | 120 [120 to 140]
Quality of muscle reaction in pronation [Median (Inter-Quartile Range); unit: units on a scale] — To grade the quality of muscle reaction according to the Modified Tardieu Scale, passive stretch is performed by taking into account the falling speed of the limb segment under gravity .The quality of muscle reaction ranges from 0 to 4. Grade 0 represents no spasticity and grade 4 represents severe spasticity. Grade 1 means slight resistance to passive stretch with no clear catch at precise angle. Grade 2 marks clear catch at precise angle followed by release. Grade 3 represents fatigable clonus occurring at precise angle, and grade 4 represents nonfatigable clonus occurring at precise angle.
  units on a scale | 2 [2 to 2]
Quality of muscle reaction in the neutral position of forearm [Median (Inter-Quartile Range); unit: units on a scale] — To grade the quality of muscle reaction according to the Modified Tardieu Scale, passive stretch is performed by taking into account the falling speed of the limb segment under gravity .The quality of muscle reaction ranges from 0 to 4. Grade 0 represents no spasticity and grade 4 represents severe spasticity. Grade 1 means slight resistance to passive stretch with no clear catch at precise angle. Grade 2 marks clear catch at precise angle followed by release. Grade 3 represents fatigable clonus occurring at precise angle, and grade 4 represents nonfatigable clonus occurring at precise angle.
  units on a scale | 2 [2 to 2]
Quality of muscle reaction in supination [Median (Inter-Quartile Range); unit: units on a scale] — To grade the quality of muscle reaction according to the Modified Tardieu Scale, passive stretch is performed by taking into account the falling speed of the limb segment under gravity .The quality of muscle reaction ranges from 0 to 4. Grade 0 represents no spasticity and grade 4 represents severe spasticity. Grade 1 means slight resistance to passive stretch with no clear catch at precise angle. Grade 2 marks clear catch at precise angle followed by release. Grade 3 represents fatigable clonus occurring at precise angle, and grade 4 represents nonfatigable clonus occurring at precise angle.
  units on a scale | 2 [2 to 2]

OUTCOME MEASURES:

1. Primary Outcome: Dynamic Component of Spasticity (Spasticity Angle)
Description: According to the Modified Tardieu Scale, the difference between the angle of slow passive motion and the angle of muscle reaction represents the dynamic component of spasticity (spasticity angle) in degree. A big difference suggests spasticity while the low difference suggests muscular contracture. In this study, dynamic component of spasticity (spasticity angle) at forearm pronation, neutral position and supination was evaluated separately.
Time Frame: 1 day (Only one measurement was performed in time (cross-sectional))
Measure: Median (Inter-Quartile Range); unit: degree
Groups:
- Spasticity Angle in Pronation: First group of three groups of paired observations consisting of participants whose measurements of dynamic component of elbow flexor spasticity were performed in the pronation position of forearm
- Spasticity Angle in Neutral Position: Second group of three groups of paired observations consisting of participants whose measurements of dynamic component of elbow flexor spasticity were performed in the neutral position of forearm
- Spasticity Angle in Supination: Third group of three groups of paired observations consisting of participants whose measurements of dynamic component of elbow flexor spasticity were performed in the supination position of forearm
Arm/Group | Spasticity Angle in Pronation | Spasticity Angle in Neutral Position | Spasticity Angle in Supination
Number analyzed (Participants) | 60 | 60 | 60
degree | 70 [50 to 80] | 60 [50 to 75] | 57.5 [30 to 70]
Statistical Analysis 1: Comparison: Spasticity Angle in Pronation vs Spasticity Angle in Neutral Position vs Spasticity Angle in Supination; Null hypothesis: no difference between dynamic components of elbow flexor spasticity (spasticity angle) in three different forearm positions. (Comparison groups were Spasticity angle in pronation, Spasticity angle in neutral position and Spasticity angle in supination); Test type: Other; p < 0.001, Friedman — p-value was adjusted for multiple comparisons. A priori threshold for statistical significance was set to 0.05/3 (0.0167)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Post-stroke Elbow Flexor Spasticity
All-Cause Mortality (participants affected / at risk) | 0/60
Serious Adverse Events (participants affected / at risk) | 0/60
Other Adverse Events (participants affected / at risk) | 0/60

LIMITATIONS AND CAVEATS:
Technical problems related to measurement in determining muscle reaction angle and slow controlled motion with a standard goniometer. The use of semi-quantitative spasticity assessment scales.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-21): https://cdn.clinicaltrials.gov/large-docs/09/NCT03563209/Prot_SAP_000.pdf